CLINICAL TRIAL: NCT03607526
Title: Barriers and Facilitators to Following the Dietary Guidelines for Vegetable Intake: Follow-up of an Intervention to Increase Vegetable Consumption
Brief Title: Barriers and Facilitators to Vegetable Intake
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC152
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Overweight; Obese
Keywords: Vegetable Intake
MeSH Terms: conditions — Overweight; Obesity | interventions — Glucose Transport Proteins, Facilitative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Barriers to Vegetable Consumption: Four groups of participants will meet for NGT sessions, identifying barriers to meeting the DGA recommendation for vegetable consumption.
  Interventions: Other: Barriers
- Facilitators to Vegetable Consumption: Four groups of participants will meet for NGT sessions, identifying facilitators to meeting the DGA recommendation for vegetable consumption.
  Interventions: Other: Facilitators

INTERVENTIONS:
Other: Barriers — NGT sessions identifying barriers to vegetable intake.
  Groups: Barriers to Vegetable Consumption
Other: Facilitators — NGT sessions identifying facilitators to vegetable intake.
  Groups: Facilitators to Vegetable Consumption

SUMMARY:
The purpose of this study is to find out why people do or do not eat vegetables.

DETAILED DESCRIPTION:
The Dietary Guidelines for Americans (DGA) stress the importance of a diet high in fruits and vegetables (FV) to achieve health benefits. Despite the recommendations, adherence is low; only 12% of the population meets the recommendation for fruits and even less of the population (9%) meets the recommendation for vegetables. Recently, it was found that vegetable consumption increased when individuals were provided the recommended daily amounts while participating in a clinical study, but returned to pre-study low levels when vegetables were no longer supplied. This result suggests that habitual consumption of FV is strongly regulated by behaviors influenced by social, environmental, and/or individual factors. Therefore, identifying regulatory factors of vegetable consumption will greatly assist in developing successful strategies to increase vegetable intake to achieve health benefits. The overall objective of this study is to examine both barriers and facilitators to adherence to consuming DGA-recommended amounts of vegetables in participants who completed a randomized controlled trial with provided vegetables or who were in a control group, using the Nominal Group Technique (NGT).

ELIGIBILITY:
Inclusion Criteria:

* Participant in NCT02585102 who gave permission to be contacted for a follow-up study.

Exclusion Criteria:

* Did not participate in NCT02585102.
* Participant in NCT02585102 who did not give permission to be contacted for a follow-up study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be limited to contacting participants who previously took part in a study (NCT02585102) and upon completion of that study indicated willingness to be contacted for a follow-up study. The original study recruited overweight or obese adults who reported consuming not more than 1 serving of vegetables per day. In that study, participants were provided vegetables or were in a control group. Research staff will send invitations to participate in one of the NGT sessions.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Barriers and facilitators to vegetable consumption | 2 hours
  NGT results providing an exhaustive list of barriers and facilitators to meeting the DGA for vegetable consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03607526/ICF_000.pdf